CLINICAL TRIAL: NCT00902863
Title: The Impact of a Course on Stress Reduction Techniques on Satisfaction, Stress, Performance, and Quality of Life in Patients With Chronic Pain
Brief Title: Impact of a Course on Stress Reduction
Acronym: YOGA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to keep patients attending yoga sessions
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. Lori Olivieri, Hamilton Health Sciences
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-070
Record Dates: First submitted 2009-05-12; First posted 2009-05-15 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Pain
Keywords: chronic pain; mindfulness; yoga; quality of life; stress
MeSH Terms: conditions — Chronic Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YOGA patients (Experimental): Patients assessed for chronic pain at our Pain Management Centre
  Interventions: Behavioral: YOGA

INTERVENTIONS:
Behavioral: YOGA — Patients with chronic pain will undergo a six week course of YOGA

SUMMARY:
This project seeks to measure the effectiveness of a course in self-management strategies (including yoga, mindfulness, and breathing exercises). The course will be provided by a certified yoga instructor to patients being followed at the Pain Management Centre, Hamilton Health Sciences (HHS).

DETAILED DESCRIPTION:
The Pain Management Centre at Hamilton Health Sciences is organizing a course in stress reduction techniques for patients with chronic pain. The Pain Centre has arranged for a local certified yoga instructor to lead a 6-week course that she has developed for our specific patient population. The course will include self-management strategies for pain control, such as breathing exercises, yoga poses, and mindfulness meditation. Standardized questionnaires and a semi-structured interview to record baseline and post-course outcomes. The study will involve the following questionnaires/surveys/interviews: 1) Canadian Occupational Performance Measure, 2) Perceived Stress Scale, 3) Burckhardt Quality of Life Scale, 4) Visual Analog Score, and 5) written questions concerning patient demographics, the patient's chronic pain condition, and their satisfaction with the course. The participants would be asked to fill out questionnaires at three different times: 1) baseline data collected within two weeks of starting course, 2) short-term outcome data within two weeks of completing course, and 3) long-term outcome data four to six months after the course.

ELIGIBILITY:
Inclusion Criteria:

* patients have a history of moderate to severe chronic pain

Exclusion Criteria:

* non-English speaking patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Performance and Satisfaction using Canadian Occupational Performance Measure (COPM) | 6 months

SECONDARY OUTCOMES:
Pain relief using VAS and pain scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Olivieri, M.D., Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Mead K, Theadom A, Byron K, Dupont S. Pilot study of a 4-week Pain Coping Strategies (PCS) programme for the chronic pain patient. Disabil Rehabil. 2007 Feb 15;29(3):199-203. doi: 10.1080/09638280600756117. PMID 17364770